CLINICAL TRIAL: NCT06331364
Title: TREATment of Lower Respiratory Tract Infection in Selected Hospitals in Southern Sri Lanka (TREAT-SL): A Stepped-wedge Cluster Randomized Trial of an Electronic Clinical Decision Support Tool (eCDST) for the Diagnosis and Treatment of Lower Respiratory Tract Infection (LRTI) in Selected Hospitals in Southern Sri Lanka
Brief Title: TREATment of Lower Respiratory Tract Infection in Selected Hospitals in Southern Sri Lanka (TREAT-SL): a Stepped-Wedge Cluster Randomized Trial
Acronym: TREAT-SL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114347; R01AI168420 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Lower Resp Tract Infection
Keywords: eCDST

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, cluster randomized, two-arm, open label
  This design combines elements of a cluster randomized trial (intervention is applied in clusters) and a before-after design (each cluster switches to intervention). All 9 pairs of wards (clusters) will start with an initial period of usual care. At intervals of 3-6 months (steps), a set of 3 pairs of wards (clusters) will switch in a randomized order to use the intervention, until all pairs of wards have crossed over. We will use the stepped-wedge design since 1) this design may provide higher statistical power, since clusters act as their own controls, 2) to reduce contamination bias, and 3) to reduce the risk of a cluster dropping out of the study if assigned to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Clinicians will be asked to use the diagnostic portion of the electronic clinical decision tool (eCDST) on their mobile phones, into which they will enter inputs and receive a diagnostic plan. Point of care (POC) testing as advised by the eCDST will be conducted by either clinical staff or trained research staff. If performed by research staff, results will be delivered on paper within 6 hours of testing to ≥ 2 primary clinicians on the team (including the consultant/ attending-level physician or senior registrar). THK, DGM, and DGH do not have an electronic medical record system. Clinicians will be asked to input the results from diagnostic testing and to follow the treatment recommendations as per the eCDST, but will be advised that the final decision regarding prescription of antimicrobials is entirely at their discretion.
  Interventions: Other: electronic clinical decision support tool (eCDST) diagnostic plan
- Usual Care Arm (No Intervention): Study staff will inform the treating clinicians to diagnose and treat patients according to usual practice. Clinicians will be able to order routine diagnostic testing as per standard practice.
  These tests may include complete blood count, chemistries, C-reactive protein (CRP) testing, erythrocyte sedimentation rate (ESR) testing, blood and sputum cultures, and chest x-ray or chest CT imaging.

INTERVENTIONS:
Other: electronic clinical decision support tool (eCDST) diagnostic plan — Participants will be followed for 30 days from enrollment to record clinical outcomes and any antimicrobials used. Analyses will compare clinical outcomes and antimicrobial use between the intervention arm and usual care.
  Arms: Intervention Arm

SUMMARY:
This is a stepped-wedge, cluster-randomized, two-arm, open-label, clinical trial of an electronic clinical decision support tool (eCDST) for the diagnosis and treatment of lower respiratory tract infection (LRTI) among patients at three sites in Southern Province, Sri Lanka.

The primary objective of this trial is to determine the impact of an electronic clinical decision support tool (eCDST) on clinical outcomes and antibacterial prescription in subjects with LRTI in the intervention group compared to the control group.

The study will enroll 765 patients ≥ 14 years of age. Medical wards will be randomized in clusters to the intervention at intervals of 3-6 months until all clusters cross over. Participants will be followed for 30 days from enrollment to record clinical outcomes and any antimicrobials prescribed (a maximum of 14 days).

ELIGIBILITY:
Inclusion Criteria:

1. Admitted within prior 48 hours
2. Have evidence of new acute respiratory illness (<14 days of symptoms), as indicated by at least one of the following:

   1. New cough or sputum production
   2. Chest pain
   3. Dyspnea or tachypnea (respiratory rate >20 breaths/minute)
   4. Abnormal lung examination
3. Have evidence of acute infection, as indicated by at least one of the following:

   1. Self-reported fever or chills
   2. Documented fever ≥38 ̊ C (100.4 ̊ F)
   3. Documented hypothermia <35.5 ̊ C (95.9 ̊ F)
   4. Leukocytosis (white blood cell count >10,000/mm3)
   5. Leukopenia (white blood cell count <3000/mm3)
   6. New altered mental status
4. Ability and willingness of patient, parent or legally authorized representative (LAR) to give informed consent
5. Ability of children 14-17 years of age to provide assent
6. Ability to complete follow-up encounter at 30 days in person or by telephone

Exclusion Criteria:

1. Hospitalized recently (within last 28 days)
2. If they have been enrolled into this clinical trial previously
3. Surgery in the past 7 days
4. If they are unable or unwilling to complete the follow-up encounter
5. If they will likely be transferred from the medical wards within 24 hours of enrollment (to another ward or to another hospital)
6. If they have underlying conditions or circumstances for which physicians would be unlikely to withhold antibacterials:

   1. Vasopressor therapy
   2. Cystic fibrosis
   3. Known severe immunosuppression (i. Cancer or another condition with neutropenia (absolute neutrophil count <1000/ microL; ii. Solid- organ or hematopoietic stem-cell transplant within the previous 90 days; iii. Active graft-versus-host disease or bronchiolitis obliterans; iv. On chronic steroids equivalent to prednisone 20mg daily for ≥ 2 weeks or other targeted cytotoxic or biologic immunosuppressants within the prior 4 weeks; v. Human immunodeficiency virus infection with a CD4 cell count <200/mm3)
   4. Have an accompanying non-respiratory infection
   5. Have evidence of a lung abscess or empyema
   6. Have respiratory failure at enrollment, evidenced by use of non-invasive or invasive ventilation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 765 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Composite of adverse outcomes that could be attributed to withholding antibacterials | Day 30
  A binary clinical endpoint consisting of a composite of adverse outcomes that could be attributed to withholding antibacterials. These outcomes would not be present at enrollment, and could occur anytime until Day 30.
Total duration of antibacterial prescription for the index visit | Index hospitalization, up to approximately 14 days
  Total duration of antibacterial prescription for the index visit will include the number of days that antibacterials are prescribed during the index hospitalization, as well as the number of days that antibacterials are prescribed at discharge from the hospital (intended use).

SECONDARY OUTCOMES:
Proportion of participants using non-invasive ventilation | Day 30
  Use of non-invasive ventilation (i.e., continuous positive airway pressure [CPAP] or bilevel positive airway pressure [BiPAP]) for treatment of the acute illness )
Proportion of participants using mechanical ventilation | Day 30
  Use of mechanical ventilation (via endotracheal tube)
Proportion of participants readmitted to the hospital | Day 30
  Proportion of participants readmitted to the hospital
Proportion of deaths | Day 30
  Proportion of deaths
Proportion of participants seeking subsequent outpatient care for the LRTI illness and receiving an antibacterial prescription | Day 30
  Proportion of participants seeking subsequent outpatient care for the LRTI illness and receiving an antibacterial prescription
Proportion of participants admitted to the intensive care unit (ICU) during index hospitalization | Index hospitalization, up to approximately 30 days
  Proportion of participants admitted to the intensive care unit (ICU) during index hospitalization
Duration of admission to the intensive care unit (ICU) during index hospitalization | Index hospitalization, up to approximately 30 days
  Duration of admission to the intensive care unit (ICU) during index hospitalization
Number of participants requiring use of supplemental oxygen by nasal cannula or face mask during index hospitalization | Index hospitalization, up to approximately 30 days
  Number of participants requiring use of supplemental oxygen by nasal cannula or face mask during index hospitalization
Duration of supplemental oxygen by nasal cannula or face mask during index hospitalization | Index hospitalization, up to approximately 30 days
  Duration of supplemental oxygen by nasal cannula or face mask during index hospitalization
Duration of non-invasive ventilation during index hospitalization | Index hospitalization, up to approximately 30 days
  Duration of non-invasive ventilation during index hospitalization
Duration of mechanical ventilation during index hospitalization | Index hospitalization, up to approximately 30 days
  Duration of mechanical ventilation during index hospitalization
Duration of index hospitalization | Index hospitalization, up to approximately 30 days
  Duration of index hospitalization
Proportion prescribed antibacterials- cumulative | Day 1, Day 2, Day 3, by discharge, and by Day 30
  Any prescription of antibacterials from enrollment to the point of assessment will be considered prescription of antibacterials.
Proportion prescribed antibacterials- at time of assessment | Day 1, Day 2, Day 3, by discharge, and by Day 30
  Prescription of antibacterials will only be assessed at the specific time of assessment
Total antibacterial exposure per patient during hospitalization | Day 30
  This is defined as the total number of days prescribed an antibacterial
Proportion prescribed oseltamivir- cumulative | Day 1, Day 2, Day 3, at discharge, and by Day 30
  Any prescription of oseltamivir from enrollment to the point of assessment will be considered prescription of oseltamivir
Proportion prescribed oseltamivir- at time of assessment | Day 1, Day 2, Day 3, at discharge, and by Day 30
  Prescription of oseltamivir will only be assessed at the specific time of assessment
Total oseltamivir exposure per patient during hospitalization | Day 30
  This is defined as the total number of days prescribed oseltamivir
Proportion prescribed SARS-CoV-2 antivirals during hospitalization- cumulative | Day 1, Day 2, Day 3, at discharge, and by Day 30
  Any prescription of SARS-CoV-2 antivirals from enrollment to the point of assessment will be considered prescription of SARS-CoV-2 antivirals
Proportion prescribed SARS-CoV-2 antivirals during hospitalization- at time of assessment | Day 1, Day 2, Day 3, at discharge, and by Day 30
  Prescription of SARS-CoV-2 antivirals will only be assessed at the specific time of assessment
Physician adherence, as measured by proportion in whom the first recommended diagnostic test (if recommended) was performed | 24 hours
  Physician adherence to the eCDST diagnostic recommendations within 24 hours of receiving recommendations, in the intervention group.
Physician adherence, as measured by the proportion in whom the second recommended diagnostic test (if recommended) was performed | 48 hours
  Physician adherence to the eCDST diagnostic recommendations within 48 hours of receiving recommendations, in the intervention group.
Physician adherence, as measured by proportion in whom the antibacterial treatment recommendation was followed | 24 hours and 48 hours
  Physician adherence, as measured by proportion in whom the antibacterial treatment recommendation was followed
Physician adherence, as measured by the proportion in whom the oseltamivir treatment recommendation was followed | 24 hours and 48 hours
  Physician adherence, as measured by the proportion in whom the oseltamivir treatment recommendation was followed
Physician adherence, as measured by the proportion in whom all treatment recommendations were followed | 24 hours and 48 hours
  Physician adherence, as measured by the proportion in whom all treatment recommendations were followed

CONTACTS AND LOCATIONS:
Overall Officials: Gayani Tillekeratne, MD, MSc, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No